CLINICAL TRIAL: NCT02179320
Title: Evaluation of the Efficacy and Neurological Effects of Dry Needling in the Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HC-GDOR-MIOFASCIAL
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2015-04

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial Pain Syndrome; Dry needling; Clinical Trial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry needling (Active Comparator): Dry needling for myofascial pain syndrome, in the trapezius muscle.
  Interventions: Procedure: Dry needling; Device: acupuncture needle 0,25 x 40mm
- Sham needling (Sham Comparator): Superficial dry needling in the trapezius muscle
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Dry needling of the painful muscles, with an acupuncture needle 0,25 x 40mm
Device: acupuncture needle 0,25 x 40mm
  Arms: Dry needling

SUMMARY:
AIM OF INVESTIGATION: To evaluate in a prospective, randomized, sham-controlled study the pattern of analgesic efficacy of trigger point dry needling in Myofascial Pain Syndrome (MPS) patients.

DETAILED DESCRIPTION:
This study will be performed in patients with shoulder pain due to excess of nociception associated with chronic Myofascial Pain Syndrome in asymmetrical unilateral trapezius muscle trigger points.

Patients will be randomly assigned to two treatment arms: Active (A) (n=20) and Sham (S) (n=21). Group A will receive actual treatment with trigger point dry needling. Group S will receive a sham treatment, with the needle inserted superficially in the skin, without reaching the muscle underneath it.

The duration and pain elicited during active and sham dry needling will be controlled for. Patients will be evaluated one week before needling (D-7), on the day of dry needling (D0) and seven days after the procedure (D+7).

Patients will fill out the Brazilian version of the Douleur Neuropathique 4, Beck Depression Inventory, Brief Pain Inventory (BPI), McGill Pain Questionnaire-SF (SFMPQ), Hospital Anxiety and Depression Scale and Global Impression of Change, and also a 14-day Carnet to more accurately evaluate their daily pain before and after the treatment.

For the evaluation of neurologic changes, we will evaluate local hyperalgesia, tactile, mechanical, static and thermal sensitivity with thermal quantitative sensorial testing (TQS), and also mapping of the painful area, before and after treatment in both D0 and D+7.

ELIGIBILITY:
Inclusion Criteria:

* Assymetric shoulder pain (VAS on painful side : VAS on non painful side > 2:1)
* Pain due to unilateral Myofascial Pain Syndrome of the trapezius muscle.
* Chronic pain, with duration of at least 3 months and VAS > 40/100
* Patients with pain at least 4 days in a week
* Patients without neurological pain, as in DN4 score less than 4
* Age over 18 years
* Patients with stable drug treatment over at least 15 days, without any acute pharmacological changes during the study
* Patients who read, understood and signed the Free and Clarified Consent Term

Exclusion Criteria:

* Patients with major depression, according to DSM-IV criteria
* History of bipolar mood disorder, panic syndrome or psychosis
* Intermittent pain history
* Refusal to sing the Consent Term
* Patients not able to attend all the follow-ups
* Patients with another pain syndrome in shoulders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Analgesic effects of dry needling | Within the first 7 days after treatment
  Maximum, average and lowest pain will be evaluated daily 7 days before the treatment, on the day of the treatment, and also 7 days after the treatment is done.

SECONDARY OUTCOMES:
Neurologic effects of dry needling | Within the first 7 days after treatment
  Tactile, mechanical, static and thermal sensitivity will be evaluated with thermal quantitative sensorial testing, as well as hyperalgesia. The painful area will also be mapped to compara before and after treatment results.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Andrade, M.D., P.h.D., Study Chair — University of Sao Paulo; Juliana T Toma, M.D., Principal Investigator — University of Sao Paulo; Irina Raicher, M.D., Principal Investigator — University of Sao Paulo; Manoel J Teixeira, M.D., P.h.D., Study Director — University of Sao Paulo; Helena H Kaziyama, M.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Yap EC. Myofascial pain--an overview. Ann Acad Med Singap. 2007 Jan;36(1):43-8. PMID 17285185
- [Background] Gerwin RD. Classification, epidemiology, and natural history of myofascial pain syndrome. Curr Pain Headache Rep. 2001 Oct;5(5):412-20. doi: 10.1007/s11916-001-0052-8. PMID 11560806
- [Background] Ga H, Choi JH, Park CH, Yoon HJ. Dry needling of trigger points with and without paraspinal needling in myofascial pain syndromes in elderly patients. J Altern Complement Med. 2007 Jul-Aug;13(6):617-24. doi: 10.1089/acm.2006.6371. PMID 17718644
- [Background] Cummings TM, White AR. Needling therapies in the management of myofascial trigger point pain: a systematic review. Arch Phys Med Rehabil. 2001 Jul;82(7):986-92. doi: 10.1053/apmr.2001.24023. PMID 11441390
- [Background] McCain GA, Bell DA, Mai FM, Halliday PD. A controlled study of the effects of a supervised cardiovascular fitness training program on the manifestations of primary fibromyalgia. Arthritis Rheum. 1988 Sep;31(9):1135-41. doi: 10.1002/art.1780310908. PMID 3048273
- [Background] Giamberardino MA. Referred muscle pain/hyperalgesia and central sensitisation. J Rehabil Med. 2003 May;(41 Suppl):85-8. doi: 10.1080/16501960310010205. PMID 12817663
- [Background] Ge HY, Fernandez-de-las-Penas C, Arendt-Nielsen L. Sympathetic facilitation of hyperalgesia evoked from myofascial tender and trigger points in patients with unilateral shoulder pain. Clin Neurophysiol. 2006 Jul;117(7):1545-50. doi: 10.1016/j.clinph.2006.03.026. Epub 2006 Jun 5. PMID 16737848
- [Background] Hong CZ, Simons DG. Pathophysiologic and electrophysiologic mechanisms of myofascial trigger points. Arch Phys Med Rehabil. 1998 Jul;79(7):863-72. doi: 10.1016/s0003-9993(98)90371-9. PMID 9685106
- [Background] Hong CZ. Treatment of myofascial pain syndrome. Curr Pain Headache Rep. 2006 Oct;10(5):345-9. doi: 10.1007/s11916-006-0058-3. PMID 16945250
- [Background] Giamberardino MA, Affaitati G, Fabrizio A, Costantini R. Myofascial pain syndromes and their evaluation. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):185-98. doi: 10.1016/j.berh.2011.01.002. PMID 22094195
- [Background] Skootsky SA, Jaeger B, Oye RK. Prevalence of myofascial pain in general internal medicine practice. West J Med. 1989 Aug;151(2):157-60. PMID 2788962
- [Background] SOLA AE, RODENBERGER ML, GETTYS BB. Incidence of hypersensitive areas in posterior shoulder muscles; a survey of two hundred young adults. Am J Phys Med. 1955 Dec;34(6):585-90. No abstract available. PMID 13268620
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Ge HY, Fernandez-de-Las-Penas C, Madeleine P, Arendt-Nielsen L. Topographical mapping and mechanical pain sensitivity of myofascial trigger points in the infraspinatus muscle. Eur J Pain. 2008 Oct;12(7):859-65. doi: 10.1016/j.ejpain.2007.12.005. Epub 2008 Jan 18. PMID 18203637